CLINICAL TRIAL: NCT02306655
Title: Coital Incontinence: Incidence and Quality of Life Impact.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University Of Perugia (Other)
Responsible Party: Principal Investigator, Antonio Luigi Pastore, MD, PhD, Assistant Professor, University of Roma La Sapienza
Other Study IDs: University of Perugia
Record Dates: First submitted 2014-11-29; First posted 2014-12-03 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Urinary Incontinence; Quality of Life; Coitus
Keywords: Coital incontinence; Incidence; quality of life
MeSH Terms: conditions — Urinary Incontinence; Coitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fundamentals of scientific research The "coital incontinence" (IC), defined as the "involuntary loss of urine in association with sexual intercourse." The incidence reported in the literature ranges from 10% to 27%, but is likely to be underestimated because of the embarrassment of the woman to report the disturbance. It was in fact estimated that only 3% of women speaks spontaneously to their doctor, and increases up to 20% only after a request by the medical staff.

The CI is traditionally divided into two forms:

1. incontinence at the time of penetration (60% of cases)
2. incontinence during orgasm (40% of cases) Many theories have been proposed to justify this form of urinary incontinence, but none has been conclusively proved .Moreover, it has not been possible, to date, to identify risk factors, anatomical or urodynamics, for this condition.

The IC is rarely a symptom isolated, but more frequently associated with other forms of urinary incontinence. In particular, the IC during penetration of associated with stress urinary incontinence (loss of urine that occurs due to coughing, sneezing and in general to all those activities that increase abdominal pressure); the IC during orgasm is associated more frequently to a condition of overactive bladder (presence of urgency, urge incontinence, increased urination day and night).

The IC has a strong impact on female sexuality and can cause loss of libido, non orgasmic, decreased sexual satisfaction and, in some cases, termination of sexual activity.

Research goals Evaluate a prospective investigation of health statistics, the incidence of coital incontinence into consideration that there are few data in the literature on this disorder and those who have reported a wide variance probably connected to how the data collection. The aim is to be able to identify a "threatening condition" which, if not evaluated, worsens the prognosis of the treatment of female urinary incontinence, a condition that has a negative impact on the quality of life of patients with significantly worse than that related to other recognized debilitating chronic diseases such as diabetes.

And this individual psychosocial cost, hardly quantifiable, must be added the cost of significant socio-economic and welfare dependents of incontinent patients, the community and national health services. It is indeed evident from international and national literature that the more incisive and determined is the strategy of information, awareness and education, and adopted much wider and earlier the diagnosis, the more significant is the socio-economic savings, as well as psycho social, we get.

Ultimate goal is to differentiate between them the two forms of incontinence coital (to penetration and during orgasm) because each of them is associated with pathogenesis and therefore to a separate treatment. And while the forms of IC penetration favorably affected the treatment of stress urinary incontinence, the forms of IC during orgasm, usually associated with a functional disorder of the detrusor (detrusor overactivity) show an inferior efficacy to treatment antimuscarinic traditionally reserved to the condition of overactive bladder and therefore need a more targeted diagnostic and individualized treatments.

Materials and methods

Self administered questionnaires will be dispensed to the patients The questionnaires,validated in Italian language, will be used, according to the guidelines of the International Consultation on Incontinence, :

* ICIQ-UI on urinary incontinence short-form: for the evaluation of symptoms and quality of life:
* Patient Perception of Bladder Condition (PPBC): to assess the impact of such a subjective condition;
* Urinary incontinence and quality of sexuality;
* Urinary incontinence and frequency of sexual activity; The questionnaire is anonymous in order to protect privacy. The patients will be recruited at the outpatient surgery and Urogynaecology urodynamics of Urology Clinic of the University of Perugia.

The investigators defined that the statistically significant number of subjects can not be less than 200 units.

The time duration of the collection of medical records was estimated at two years.

There are no extremes of the conflict of interest, will not be tested or used drugs or medical equipment.

ELIGIBILITY:
Inclusion Criteria:

Female patients with age > 18 y.o. Stable relationship for at least 6 months At least one sexual intercourse every 2 weeks

Exclusion Criteria:

Male patients Female patients aged < 18 y.o. Patients without a stable relationship or with no sexual activity (as defined for at least one sexual intercourse every 2 weeks)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with sexual activity and with stable relationship for at least six months
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-11 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life evaluation in patients with coital incontinence | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Urology Unit, Sapienza University of Rome, Latina
  - Urogynecology Unit, Urology Clinic, University of Perugia, Perugia